CLINICAL TRIAL: NCT00840268
Title: A Study of Hydroxypropyl Guar Galactomannan 0.25% (HPGG) Versus Vehicle in Dry Eye Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-34
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Dry Eye
Keywords: OSDI; corneal staining; Dry Eye; Dry Eye Signs and Symptoms in Dry Eye Patients
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPGG 0.25% (Experimental): Hydroxypropyl Guar Galactomannan (HPGG) 0.25% ophthalmic gel, 1 drop per eye twice daily (BID) (in the morning upon awakening and in the evening prior to bedtime) for 21 days (Treatment phase).
  Interventions: Drug: Hydroxypropyl Guar Galactomannan (HPGG) 0.25% ophthalmic gel
- HPGG Vehicle (Placebo Comparator): Hydroxypropyl Guar Galactomannan Vehicle, 1 drop per eye twice daily (BID) (in the morning upon awakening and in the evening prior to bedtime) for 21 days (Treatment phase).
  Interventions: Drug: Hydroxypropyl Guar Galactomannan Vehicle

INTERVENTIONS:
Drug: Hydroxypropyl Guar Galactomannan (HPGG) 0.25% ophthalmic gel
  Other Names: HPGG
  Arms: HPGG 0.25%
Drug: Hydroxypropyl Guar Galactomannan Vehicle — Inactive ingredients used as a placebo comparator
  Other Names: HPGG Vehicle
  Arms: HPGG Vehicle

SUMMARY:
The purpose of this study is to demonstrate efficacy of Hydroxypropyl Guar Galactomannan 0.25% (HPGG) ophthalmic gel compared to Vehicle for the treatment of dry eye.

DETAILED DESCRIPTION:
A 7-day Vehicle pre-randomization (run-in) phase during which all patients will receive 1 drop of Vehicle in each eye twice daily will precede the 21-day treatment phase, for an overall study duration of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Must read, sign, and date an informed consent document and HIPAA privacy document.
* Diagnosis of dry eye at Visit 1 (Day 0).
* Able and willing to follow study instructions.
* Best corrected visual acuity (BCVA) of 0.6 logMAR or better in each eye as assessed using an ETDRS chart at Visit 1.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Diagnosis of Sjogren's syndrome (or suspected to have Sjogren's syndrome).
* History or evidence of ocular or intraocular surgery in either eye within the previous year.
* History or evidence of serious ocular trauma in either eye within the previous 6 months.
* History or evidence of corneal transplant or transplant variant procedures.
* History of intolerance or hypersensitivity to any component of the study medications.
* History of glaucoma or current ocular hypertension in either eye, or treatment for either condition within 6 months prior to Visit 1.
* History or evidence of corneal conditions, other than dry eye, that may affect the corneal structure.
* Use of any concomitant topical ocular medications including artificial tears during the study period.
* Females of childbearing potential if breastfeeding, unwilling to undergo urine pregnancy test at screening and upon exiting the study, have a positive urine pregnancy test at screening, intend to become pregnant during the study, or do not agree to use adequate birth control methods for the duration of the study.
* Use of RESTASIS® 0.05% or an ocular steroid within 30 days of Visit 1.
* Use of systemic medications that have not been stable for 30 days prior to Visit 1.
* Any ocular condition that may preclude the safe administration of the test article.
* Unwilling to discontinue contact lens wear at least 4 weeks prior to Visit 1, and during the study period.
* Use of punctal plugs or punctal cautery.
* Use of lid scrubs/warm compresses within 14 days of Visit 1.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in sodium fluorescein corneal staining score | Baseline (Day 7), Up to Day 28

SECONDARY OUTCOMES:
Mean change from baseline in Dry Eye Symptom Questionnaire (OSDI) score | Baseline (Day 7), Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jay H. Mashburn, Study Director — Alcon Research